CLINICAL TRIAL: NCT06807333
Title: Transforming Diabetes Care: Pharmacist-Led Education and Its Impact on Patient Knowledge, Self-Management, and Health Outcomes
Acronym: TRIPLE-CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa International Hospital (Other)
Responsible Party: Principal Investigator, SARA YAHYA, Principal Pharmacist, Shifa International Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 318-24
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
Keywords: Pharmacist; Patient Knowledge; Self-Management; Health Outcome; HbA1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: Participants will be entertained as part of their regular appointment for prescription filling without any information of which group they are assigned in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Group (Experimental): Lifestyle Modifications: Education on healthy meal choices and physical activity to support diabetes management. Disease Education: In-depth information on diabetes, blood sugar control, and the prevention of complications. Self-Management Tools: Provision of blood glucose monitoring charts and practical strategies for daily diabetes care. Counseling: Personalized counseling to address emotional aspects, stress management, and confidence in managing diabetes.
  Interventions: Behavioral: Pharmacist led Education

INTERVENTIONS:
Behavioral: Pharmacist led Education — Pharmacist-led education for diabetic patients focuses on enhancing their understanding of the disease, improving self-management skills, and promoting better health outcomes. The education covers key aspects of diabetes, such as the importance of blood sugar control, the role of diet and exercise, and how to monitor blood glucose levels. Patients are also taught effective self-management strategies, including how to make healthy food choices, incorporate physical activity into daily routines, and manage potential complications. By providing tailored education, pharmacists aim to empower patients to take an active role in their care, which can lead to improved disease management, better glycemic control, and reduced risk of complications.

SUMMARY:
This interventional study is to evaluate the impact of pharmacist-led education on diabetic patients' knowledge, self-management, and overall health outcomes. Participants in this study will attend pharmacist-led educational sessions designed to improve their understanding of diabetes and self-care practices. Researchers will assess changes in patients' knowledge, self-management behaviors, and clinical health markers before and after the intervention. The study will compare pre- and post-intervention results to determine the effectiveness of pharmacist-led education in transforming diabetes care.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether pharmacist-led education can enhance the knowledge, self-management behaviors, and health outcomes of diabetic patients. Effective diabetes management requires a comprehensive understanding of the disease, adherence to lifestyle modifications, and consistent monitoring of health indicators. Poor knowledge and suboptimal self-care can lead to inadequate glycemic control, complications, and reduced quality of life. This study will evaluate the impact of pharmacist-led educational interventions on patients' motivation, diabetes-related knowledge, and self-care behaviors, as well as their effects on clinical outcomes, including improved HbA1c levels, reduced hypo- and hyperglycemic episodes, and enhanced patient satisfaction. By addressing these critical aspects, the study aims to highlight the transformative role of pharmacist-led education in advancing diabetes care and fostering sustainable, patient-centered healthcare practices.

ELIGIBILITY:
Inclusion Criteria:

* We will include all confirmed diabetic patients who visit the SIH endocrinology OPD Clinic during the study duration.

  * Both male and female patients visiting the Endocrinology Unit of the hospital will be eligible.
  * Patients with HbA1c levels greater than 8% will be included.
  * Both follow-up and newly diagnosed patients will be considered.
  * Patients who sign the informed consent form will be enrolled in the study.

Exclusion Criteria:

* We will exclude patients with gestational diabetes mellitus (GDM).

  * Patients with central obesity will not be included in the study.
  * Type 1 diabetes mellitus (DM) patients under the age of 20 will be excluded.
  * Patients with inadequate medical history will be excluded from participation.
  * Patients with HbA1c levels less than 8% will not be included.
  * Patients who do not provide informed consent or express a lack of interest in the study will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 385 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes Knowledge Score(DKQ-24) | 3 months
  Patient's diabetes knowledge will be assessed using the Diabetes Knowledge Questionnaire (DKQ). The DKQ is a tool used to evaluate a patient's understanding of diabetes, including aspects such as blood sugar control, diet, exercise, and medication management. It consists of close-ended questions, with scores ranging from 0 to 100, where a higher score indicates a better level of knowledge regarding diabetes management.
Diabetes Management Self-Efficacy Score (DMSQ-16) | 3 months
  Patient's diabetes self-management will be assessed using the Diabetes Self-Management Questionnaire (DMSQ). The DMSQ is a tool used to evaluate a patient's ability to manage their diabetes through self-care practices, including diet, physical activity, blood sugar monitoring, and medication adherence. It consists of close-ended questions, with scores ranging from 0 to 100, where a higher score reflects better self-management behaviors in managing diabetes.
HbA1C Levels (%) | 3 months
  Patient's health outcomes will be assessed using HbA1c levels. HbA1c (glycated hemoglobin) is a blood test used to measure a patient's average blood sugar level over the past 3 months. It is a key indicator of diabetes management and glycemic control. The HbA1c level is reported as a percentage, with lower percentages indicating better control of blood sugar. A target HbA1c level of less than 7% is typically recommended for most diabetic patients. The score can range from high percentages (indicating poor control) to lower percentages (indicating better glycemic control).

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Farooq, Mphil, Study Director — Shifa International Hospital; Sara Ghulam Yahya, Ms., Principal Investigator — Shifa International Hospital; Faiza Abbas, Pharm-D, Study Chair — Shifa International Hospital; Matti Ullah, PhD, Study Chair — Hamdard University Islamabad Campus; Salwa Ahsan, Study Chair — Shifa International Hospital; Osama Ishtiaq, Endocrinologist, Study Chair — Shifa International Hospital
Locations (1):
- Shifa International Hospital, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided